CLINICAL TRIAL: NCT02434770
Title: A Phase III Single-blind, Randomized, Controlled Study in Healthy Kenyan Infants to Assess the Immunogenicity and Safety of Beijing TiantanBio Liquid Bivalent Oral Poliomyelitis Vaccine (bOPV) in Comparison to a WHO Prequalified Comparator bOPV
Brief Title: Immunogenicity and Safety of Liquid Bivalent Oral Poliomyelitis Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Beijing Bio-Institute Biological Products Co., Ltd., formerly Beijing TiantanBio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VAC-015
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- BBIBP bOPV Lot 1 (Experimental): Infants received 2 drops of liquid bivalent oral polio vaccine (bOPV) manufactured by BBIBP, Lot 1, administered directly into the mouth in the first two weeks of life, and at 6, 10, and 14 weeks of age.
  Interventions: Biological: BBIBP Bivalent Oral Poliomyelitis Vaccine Lot 1
- BBIBP bOPV Lot 2 (Experimental): Infants received 2 drops of liquid bivalent oral polio vaccine (bOPV) manufactured by BBIBP, Lot 2, administered directly into the mouth in the first two weeks of life, and at 6, 10, and 14 weeks of age.
  Interventions: Biological: BBIBP Bivalent Oral Poliomyelitis Vaccine Lot 2
- BioFarma bOPV (Active Comparator): Infants received 2 drops of WHO prequalified liquid bivalent oral polio vaccine manufactured by BioFarma, administered directly into the mouth in the first two weeks of life, and at 6, 10, and 14 weeks of age.
  Interventions: Biological: BioFarma Bivalent Oral Poliomyelitis Vaccine

INTERVENTIONS:
Biological: BBIBP Bivalent Oral Poliomyelitis Vaccine Lot 1 — Each dose of bOPV (2 drops, 0.1 ml) contains attenuated Sabin strains of poliovirus serotypes 1 and 3, with at least 10^6 cell culture infectious dose 50% (CCID50)/dose and 10^5.8 CCID50/dose, respectively.
  Other Names: Poliomyelitis (Live) Vaccine Type I Type III (Human Diploid Cell), Oral
  Arms: BBIBP bOPV Lot 1
Biological: BBIBP Bivalent Oral Poliomyelitis Vaccine Lot 2 — Each dose of bOPV (2 drops, 0.1 ml) contains types 1 and 3 attenuated polioviruses (Sabin), with at least 10^6 CCID50/dose and 10^5.8 CCID50/dose, respectively.
  Other Names: Poliomyelitis (Live) Vaccine Type I Type III (Human Diploid Cell), Oral
  Arms: BBIBP bOPV Lot 2
Biological: BioFarma Bivalent Oral Poliomyelitis Vaccine — Each dose of the WHO prequalified Bio Farma bOPV (2 drops, 0.1 ml) contains attenuated Sabin strains of poliovirus serotypes 1 and 3, with at least 10^6 and 10^5.8 infective units per dose, respectively.
  Arms: BioFarma bOPV

SUMMARY:
The purpose of this study will be to evaluate whether a bivalent oral polio vaccine (bOPV) manufactured by Beijing Bio-Institute Biological Products Co., Ltd (BBIBP) has a similar immunogenicity profile to a WHO prequalified bOPV.

DETAILED DESCRIPTION:
BBIBP has been one of the two suppliers of trivalent oral polio vaccine (tOPV) in China since 1985, with control of polio in China evidence of the effectiveness of its vaccine. The company plans to introduce a liquid formulation of bOPV (types 1 and 3) to meet increasing global demand with the phasing-out of tOPV. The proposed study is intended to provide data sufficient to obtain World Heath Organization (WHO) prequalification for the BBIBP bOPV, thus making the vaccine available to help meet global demand.

Infants were enrolled and randomized prior to the birth dose of bOPV. The first dose of study vaccine was administered during the first two weeks of life and then co-administered with the primary Expanded Programme on Immunization (EPI) series vaccines in Kenya at 6, 10 and 14 weeks of age. The Kenya EPI schedule includes the following additional vaccines:

* Bacille Calmette-Guérin Vaccine (BCG) at birth
* Diphtheria and Tetanus Toxoid with Whole Cell Pertussis, Haemophilus influenzae Type V vaccine (Hib), and Hepatitis B Vaccine (DTwPHibHep) at 6, 10, 14 weeks;
* Pneumococcal Conjugate vaccine (PCV) at 6, 10, 14 weeks
* Rotavirus vaccine (Rotarix) at 6, 10 weeks

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full-term infants, as established by medical history and clinical examination before entering into the study.
* Parents willing to provide written informed consent.
* Age: infants less than 2 weeks of age at the time of enrollment (from the 1st through the 14th day of life, inclusive)

Exclusion Criteria:

* Birth weight (as documented at first medical contact) less than 2.5 kg
* Presence of diarrhea or vomiting in the previous 24 hours or on the day of enrollment (temporary exclusion)
* Presence of fever (> 37.5°C) on the day of enrollment (temporary exclusion)
* Acute disease at the time of enrollment (temporary exclusion)
* Significant malnutrition as per Investigator's judgment
* Concurrent participation in another clinical study at any time during the study period in which the infant will be exposed to an investigational or a non-investigational product
* Presence of any significant systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the child's health or is likely to result in non-conformance to the protocol
* Known or suspected impairment of immunological function (including human immunodeficiency virus [HIV] exposure) based on medical history and physical examination
* Previous receipt of polio virus vaccine
* Household contact with a known immunosuppressed individual
* Unwillingness or inability of parents for active follow-up by the study staff
* History of any neurological disorders or seizures
* Any medical condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence or a participant's ability to give informed consent
* Maternal HIV infection

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cowden, MD, MSPH, Study Chair — US Army Medical Research Unit-Kenya
Locations (2):
- Kenya (2):
  - Kenya Medical Research Institute/Walter Reed Project, Kisumu, Nyanza
  - Kenya Medical Research Institute (KEMRI)/Walter Reed Project, Kericho

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the communities in the vicinity of the study clinics (KEMRI/Walter Reed Project Kombewa Clinical Research Center and Obama Children's Hospital in Kisumu and at the Kenya Medical Research Institute/Walter Reed Project in Kericho, Kenya).
Pre-assignment Details: Infants were enrolled prior to receipt of the birth dose of bivalent oral poliomyelitis vaccine (bOPV} and were were allocated to 1 of 3 arms:
  1. Beijing Bio-Institute Biological Products Co., Ltd. (BBIBP) liquid bOPV Lot 1;
  2. BBIBP liquid bOPV Lot 2; and
  3. World Health Organization (WHO) prequalified comparator bOPV (BioFarma).
Period: Week 1 to Week 18
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV
Started | 250 | 250 | 250
Received at Least One Vaccination | 249 | 250 | 250
Completed | 235 | 228 | 233
Not Completed | 15 | 22 | 17
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 6 | 12 | 5
Not completed — Received Non-study Polio Vaccine | 8 | 10 | 9
Not completed — Relocated Out of Study Area | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Period: Week 18 to Week
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV
Started | 235 | 228 | 233
Completed | 227 | 220 | 227
Not Completed | 8 | 8 | 6
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Received Non-study Polio Vaccine | 6 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV | Total
Number analyzed (Participants) | 249 | 250 | 250 | 749
Age, Continuous [Median (Full Range); unit: days] | 1.0 [0 to 14] | 1.0 [0 to 13] | 1.0 [0 to 14] | 1.0 [0 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 111 | 121 | 355
  Male | 126 | 139 | 129 | 394
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 248 | 250 | 250 | 748
  White | 0 | 0 | 0 | 0
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 249 | 250 | 250 | 749
Length at Enrollment [Median (Full Range); unit: centimeters] | 49.5 [45.0 to 55.0] | 49.5 [44.0 to 62.0] | 49.0 [37.0 to 54.5] | 49.5 [37.0 to 62.0]
Weight at Enrollment [Median (Full Range); unit: kilograms] | 3.2 [2.4 to 4.5] | 3.1 [2.4 to 4.5] | 3.1 [2.3 to 4.9] | 3.1 [2.3 to 4.9]
Body Mass Index (BMI) at Enrollment [Median (Full Range); unit: kg/m^2] | 12.9 [9.9 to 18.0] | 13.0 [8.1 to 17.5] | 12.8 [10.0 to 25.6] | 12.9 [8.1 to 25.6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any Systemic Reactogenicity, by Maximum Severity
Description: Solicited systemic reactogenicity events evaluated during the week after each vaccination included fever, vomiting, diarrhea, decreased appetite/ poor feeding, irritability, and decreased activity. Reactions were recorded by participant's parents via memory aid. Each event was graded as:
  Mild (Grade 1): No or minimal interference with usual activities; no medical intervention/therapy required, Moderate (Grade 2): Greater than minimal interference with usual activities; no or minimal medical intervention/therapy required, Severe (Grade 3): Marked limitation in ability to perform usual activities; medical intervention/therapy required, or Potentially life-threatening (Grade 4): Inability to perform basic functions OR Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
  The overall number of participants who experienced any systemic reaction is reported. Grades are based on maximum severity per participant.
Time Frame: 7 days after each vaccination (Weeks 0, 6, 10, and 14)
Population: The safety population included all enrolled participants who had safety data available, assigned according to the actual treatment received at Day 0.
Measure: Count of Participants; unit: Participants
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 249 | 250 | 250
Participants
  Any systemic reaction | 187 | 179 | 175
  Grade 1 | 149 | 139 | 153
  Grade 2 | 32 | 32 | 18
  Grade 3 | 6 | 8 | 4

2. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Adverse events were graded as mild (Grade 1 = No or minimal interference with usual activities; no medical intervention/therapy required), moderate (Grade 2 = Greater than minimal interference with usual activities; no or minimal medical intervention/therapy required), severe (Grade 3 = Marked limitation in ability to perform usual activities; medical intervention/therapy required), or potentially life-threatening (Grade 4 = Inability to perform basic functions OR Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death).
  The overall number of participants who experienced any adverse event is reported. Grades are based on maximum severity per participant.
Time Frame: From the time of the first vaccination through 28 days after each vaccination (up to Day 126).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 249 | 250 | 250
Participants
  Any adverse event | 143 | 142 | 151
  Grade 1 | 111 | 114 | 117
  Grade 2 | 24 | 17 | 27
  Grade 3 | 7 | 10 | 7
  Grade 4 | 0 | 1 | 0
  Death | 1 | 0 | 0

3. Primary Outcome: Anti-polio Neutralizing Antibody Geometric Mean Titers (GMT): Serotype 1
Description: The assays for determination of anti-poliovirus neutralizing antibodies at the National Institutes for Food and Drug Control (NIFDC) were validated.
  Anti-polio antibody titer four weeks after the fourth vaccination was adjusted for the decrease in maternal antibodies based on a half-life of 28 days.
Time Frame: Screening and 4 weeks post vaccination 4 (Week 18)
Population: Per Protocol Immunogenicity (PP-IMM) population includes all enrolled participants who were randomized, received all 4 doses of bOPV per the assigned treatment group, had post-vaccination immunogenicity measurement(s),and no major protocol violations that would have potentially interfered with the immunogenicity assessment of the study vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- BBIBP bOPV Lot 1 + Lot 2: Infants received 2 drops of liquid bivalent oral polio vaccine (bOPV) manufactured by BBIBP, Lot 1 or Lot 2, administered directly into the mouth in the first two weeks of life, and at 6, 10, and 14 weeks of age.
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 226 | 217 | 443 | 225
titer
  Screening | 40.9 [33.7 to 49.7] | 41.5 [34.0 to 50.6] | 41.2 [35.9 to 47.3] | 47.7 [38.4 to 59.3]
  4 Weeks after vaccination 4 | 55192 [45821 to 66478] | 65790 [55728 to 77668] | 60151 [53095 to 68144] | 55634 [46484 to 66586]
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 vs BBIBP bOPV Lot 2; Test type: Equivalence — Primary efficacy objective 1 of this study was to demonstrate the equivalence of two lots of BBIBP bOPV in terms of post-vaccination anti-polio neutralizing antibody GMTs. The immune response of the two lots of BBIBP bOPV would be declared equivalent if the 95% confidence interval (CI) for the serotype-specific GMT ratio for both serotypes was contained within (0.5, 2.0); Ratio of Geometric Mean Titers = 0.84, 95% CI 2-sided [0.65 to 1.08] — Lot 1 / Lot 2
Statistical Analysis 2: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; Test type: Non-Inferiority — Secondary efficacy objective 2 of this study was to demonstrate the non-inferiority of the two lots of BBIBP bOPV combined to the WHO control in terms of post-vaccination anti-polio neutralizing antibody GMTs. The two Lots combined would be declared non-inferior to the WHO control if the lower limit of the 95% CI for the serotype-specific GMT ratio of BBIBP Lots 1+2 over WHO control for both serotypes was > 0.5; Ratio of Geometric Mean Titers = 1.08, 95% CI 2-sided [0.87 to 1.34] — Lot 1 + Lot 2 / BioFarma bOPV

4. Primary Outcome: Anti-polio Neutralizing Antibody Geometric Mean Titers: Serotype 3
Description: as for outcome 3
Time Frame: Screening and 4 weeks post vaccination 4 (Week 18)
Population: Per Protocol Immunogenicity (PP-IMM) population
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 226 | 217 | 443 | 225
titer
  Screening | 12.5 [10.7 to 14.6] | 15.6 [12.8 to 19.0] | 13.9 [12.3 to 15.8] | 14.3 [12.0 to 17.1]
  4 Weeks after vaccination 4 | 11374 [9686 to 13355] | 12390 [10559 to 14539] | 11861 [10594 to 13280] | 8063 [6811 to 9545]
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 vs BBIBP bOPV Lot 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of Geometric Mean Titers = 0.92, 95% CI 2-sided [0.73 to 1.15] — Lot 1 / Lot 2
Statistical Analysis 2: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Ratio of Geometric Mean Titers = 1.47, 95% CI 2-sided [1.21 to 1.79] — BBIBP bOPV Lot 1 + Lot 2 / BioFarma bOPV

5. Primary Outcome: Number of Infants With Serotype-specific Anti-polio Neutralizing Antibody Seroconversion 4 Weeks After Last Dose
Description: The assays for determination of anti-poliovirus neutralizing antibodies at the National Institutes for Food and Drug Control (NIFDC) were validated.
  Seroconversion was defined as a titer ≥ 1:8 if seronegative at screening, otherwise a ≥ 4-fold increase in adjusted titers (i.e., adjusted for the decay in maternal antibodies, based on a half life of 28 days).
Time Frame: 4 weeks post vaccination 4 (Week 18)
Population: Per Protocol Immunogenicity (PP-IMM) population
Measure: Count of Participants; unit: Participants
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 226 | 217 | 443 | 225
Participants
  Serotype 1 | 223 | 215 | 438 | 219
  Serotype 3 | 223 | 214 | 437 | 217
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; For serotype 1; Test type: Non-Inferiority — Primary efficacy objective 2 of this study was to demonstrate the non-inferiority of the two lots of BBIBP bOPV combined to the WHO control in terms of post-vaccination anti-polio neutralizing antibody seroconversion rates. The immune response of the combined lots of BBIBP bOPV would be declared non-inferior to the WHO control if the lower limit of the 95% CI for the difference in percent responders is greater than negative 10, provided the two lots are declared equivalent; Difference in seroconversion rate = 1.5, 95% CI 2-sided [-0.5 to 4.6] — BBIBP bOPV (Lot 1 + Lot 2) - BioFarma bOPV
Statistical Analysis 2: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; For Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Difference in seroconversion rate = 2.2, 95% CI 2-sided [-0.1 to 5.6] — BBIBP bOPV (Lot 1 + Lot 2) - BioFarma bOPV
Statistical Analysis 3: Comparison: BBIBP bOPV Lot 1 vs BBIBP bOPV Lot 2; For Serotype 1; Test type: Other — Secondary efficacy objective 1 of this study was to show consistency of the two lots in terms of post-vaccination anti-polio neutralizing antibody seroconversion rates. The two lots would be declared consistent if the upper and lower limits of the 95% CI for the difference in seroconversion rates is within 10 percentage points of the observed difference for both serotypes; Difference in seroconversion rate = -0.4, 95% CI 2-sided [-3.0 to 2.1] — Lot 1 - Lot 2
Statistical Analysis 4: Comparison: BBIBP bOPV Lot 1 vs BBIBP bOPV Lot 2; For Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 3]; Difference in seroconversion rate = 0.1, 95% CI 2-sided [-2.6 to 2.8] — Lot 1 - Lot 2

6. Secondary Outcome: Anti-hepatitis B Surface Antigen (HBsAg) Geometric Mean Titers
Description: Anti-HBsAg titers were measured to assess the impact of concomitant administration of BBIBP liquid bOPV on immune responses to other Expanded Programme on Immunization (EPI) vaccines in comparison to that of the WHO pre-qualified bOPV, 4 weeks after the fourth vaccination.
  The enzyme-linked immunosorbent assay (ELISA) assays for serum antibodies to HBsAg were performed at the Children's Hospital Medical Center (CCHMC). The HBsAb assay was a qualified assay using a kit from BioRad.
Time Frame: 4 weeks post vaccination 4 (Week 18)
Population: Participants who received all 4 bOPV vaccinations and ≥ 3 hepatitis B virus vaccinations at least 21 days prior to blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 209 | 203 | 412 | 209
titer | 320 [246 to 416] | 322 [255 to 407] | 321 [269 to 383] | 267 [207 to 345]
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; Test type: Non-Inferiority — To show non-inferiority of Lots 1+2 combined versus BioFarma bOPV Control, the lower limit of the 95% CI must be > 0.5; Ratio of Geometric Mean Titers = 1.20, 95% CI 2-sided [0.89 to 1.63] — Lot 1 + Lot 2 / BioFarma bOPV

7. Secondary Outcome: Number of Infants With Anti-hepatitis B Surface Antigen (HBsAg) Seroprotection
Description: Seroprotection was defined as a HBsAg titer ≥ 1:10 The ELISA assays for serum antibodies to HBsAg were performed at the Children's Hospital Medical Center (CCHMC). The HBsAb assay was a qualified assay using a kit from BioRad.
Time Frame: 28 days after vaccination 4
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 209 | 203 | 412 | 209
Participants | 192 | 194 | 386 | 196
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; Test type: Other; p = 0.5586, Fisher's exact 1-tailed test; Fisher's exact 1-tailed test of a lower rate in Lots 1+2; Difference in seroprotection rate = -0.09, 95% CI 2-sided [-3.86 to 4.48] — BBIBP bOPV (Lot 1 + Lot 2) - BioFarma bOPV

8. Secondary Outcome: Anti-Rotavirus Immunoglobulin A (IgA) Geometric Mean Titers
Description: Anti-rotavirus immunoglobulin A titers were measured to assess the impact of concomitant administration of BBIBP liquid bOPV on immune responses to other Expanded Programme on Immunization (EPI) vaccines in comparison to that of the WHO pre-qualified bOPV, 4 weeks after the fourth vaccination.
  The ELISA assay for antibodies to rotavirus was performed at the Children's Hospital Medical Center (CCHMC) using a validated in-house assay.
Time Frame: 4 weeks post vaccination 4 (Week 18)
Population: Participants who received all 4 bOPV vaccinations and ≥ 2 Rotavirus vaccinations at least 21 days prior to blood draw
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BBIBP bOPV Lot 1 + Lot 2 | BioFarma bOPV
Number analyzed (Participants) | 223 | 206 | 429 | 220
titer | 22.7 [17.6 to 29.6] | 35.8 [26.8 to 47.8] | 28.3 [23.3 to 34.2] | 28.6 [21.5 to 37.9]
Statistical Analysis 1: Comparison: BBIBP bOPV Lot 1 + Lot 2 vs BioFarma bOPV; Test type: Non-Inferiority — To show non-inferiority of Lots 1+2 combined versus BioFarma bOPV Control, the lower limit of the 95% CI must be > 0.5; Ratio of Geometric Mean Titers = 0.99, 95% CI 2-sided [0.71 to 1.38] — Lot 1 + Lot 2 / BioFarma bOPV

ADVERSE EVENTS:
Time Frame: From the time of the first vaccination through completion of the study at 3 months after the last vaccination (Day 182) for serious adverse events and through 28 days after each vaccination (up to Day 126) for non-serious adverse events.
Arm/Group | BBIBP bOPV Lot 1 | BBIBP bOPV Lot 2 | BioFarma bOPV
All-Cause Mortality (participants affected / at risk) | 1/249 | 0/250 | 0/250
Serious Adverse Events (participants affected / at risk) | 13/249 | 16/250 | 17/250
Other Adverse Events (participants affected / at risk) | 143/249 | 142/250 | 151/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBIBP bOPV Lot 1 (N=249) | BBIBP bOPV Lot 2 (N=250) | BioFarma bOPV (N=250)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Breast abcess (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Malaria (Infections and infestations) | 0 | 2 | 2
Meningitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 7 | 6
Pyomyositis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sepsis neonatal (Infections and infestations) | 4 | 2 | 5
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Convulsion neonatal (Nervous system disorders) | 0 | 0 | 1
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 3 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Herbal toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBIBP bOPV Lot 1 (N=249) | BBIBP bOPV Lot 2 (N=250) | BioFarma bOPV (N=250)
Anaemia (Blood and lymphatic system disorders) | 6 | 13 | 19
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 1 | 1
Hydrocele (Congenital, familial and genetic disorders) | 3 | 3 | 2
Laryngomalacia (Congenital, familial and genetic disorders) | 1 | 3 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 50 | 51 | 51
Anal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 31 | 31 | 26
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 2 | 5 | 5
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gingival discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Gingival disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pruritus (Gastrointestinal disorders) | 0 | 0 | 1
Infantile colic (Gastrointestinal disorders) | 1 | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 6 | 4 | 7
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Abscess sterile (General disorders) | 2 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0
Developmental delay (General disorders) | 0 | 1 | 0
Granuloma (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 5 | 2
Injection site swelling (General disorders) | 2 | 1 | 1
Irritability postvaccinal (General disorders) | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 13 | 12 | 9
Swelling (General disorders) | 1 | 1 | 0
Vaccination site pain (for other EPI vaccines) (General disorders) | 0 | 1 | 0
Vaccination site swelling (for other EPI vaccines) (General disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 2 | 2
Abscess (Infections and infestations) | 4 | 4 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 1
Body tinea (Infections and infestations) | 2 | 2 | 3
Bronchiolitis (Infections and infestations) | 2 | 0 | 1
Conjunctivitis (Infections and infestations) | 36 | 32 | 30
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 4
Dysentery (Infections and infestations) | 0 | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Eye infection bacterial (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 4 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 19 | 7 | 16
Impetigo (Infections and infestations) | 11 | 8 | 6
Malaria (Infections and infestations) | 10 | 10 | 12
Mastitis (Infections and infestations) | 0 | 0 | 1
Myiasis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3
Omphalitis (Infections and infestations) | 8 | 4 | 8
Ophthalmia neonatorum (Infections and infestations) | 5 | 8 | 1
Oral candidiasis (Infections and infestations) | 8 | 13 | 8
Otitis media (Infections and infestations) | 2 | 0 | 2
Otitis media acute (Infections and infestations) | 2 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 6
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 4
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 7 | 5 | 5
Sepsis neonatal (Infections and infestations) | 3 | 5 | 5
Septic rash (Infections and infestations) | 17 | 22 | 17
Skin bacterial infection (Infections and infestations) | 1 | 3 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 1
Tinea capitis (Infections and infestations) | 4 | 1 | 1
Tinea faciei (Infections and infestations) | 2 | 1 | 2
Tinea infection (Infections and infestations) | 0 | 0 | 1
Umbilical sepsis (Infections and infestations) | 2 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 109 | 95 | 100
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Varicella (Infections and infestations) | 2 | 1 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 6 | 4 | 6
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Umbilical cord haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 1
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 8 | 6 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 4 | 3
Eczema (Skin and subcutaneous tissue disorders) | 8 | 15 | 13
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 11 | 10 | 8
Miliaria (Skin and subcutaneous tissue disorders) | 43 | 45 | 42
Rash (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5 | 12
Rash papular (Skin and subcutaneous tissue disorders) | 20 | 16 | 24
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Umbilical haematoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No